CLINICAL TRIAL: NCT04990843
Title: E-Drone: Transforming the Energy Demand of Supply Chains Through Integrated UAV-to-land Logistics for 2030
Acronym: E-Drone
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: University of Southampton (Other); University College, London (Other); University of Leeds (Other)
Responsible Party: Sponsor
Other Study IDs: RED 11731; 295372 (Other: IRAS); EP/V002619/1 (Other Grant/Funding Number: The Engineering and Physical Sciences Research Council)
Record Dates: First submitted 2021-07-15; First posted 2021-08-05 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Un-crewed aerial vehicles; Integrated logistics; Healthcare; Energy demand; Social practices; Governance
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vans are the fastest-growing category of licensed road vehicle in the UK with growing carbon dioxide (CO2) emissions. The proposed research into how Unmanned Aerial Vehicles (UAVs) and land logistics systems can be combined and managed will provide fundamental new understanding into the impacts of regulation and operating criteria on energy efficiency and costs. Medical logistics could be the first domain to utilise UAVs on a commercial scale, with preliminary analysis on pathology logistics within Southampton indicating that UAVs would significantly reduce CO2 emissions. With the National Health Service (NHS) spending an estimated £2.5 billion annually on pathology logistics and with patient numbers rising, there is a need to re-think how logistics costs could be reduced whilst improving bleed-to-diagnosis times for patients and energy demand.

The research vision is to examine the energy reduction potential of logistics solutions involving UAVs operating alongside sustainable last-mile delivery solutions (cargo cycles and walking porters via micro-consolidation points).

This involves understanding UAV operations in airspace shared with manned aircraft. The project focuses on a case study and trials based around NHS pathology sample transportation in the Solent and Dorset region. The key research objectives are to:

1. Investigate the collective transport and energy impacts of current 'business-as-usual' NHS pathology logistics across the Solent region;
2. Develop new simulation tools to quantify the energy consumption of UAVs and land logistics systems resulting from new types of traffic regulation for shared airspace and the operating requirements of UAVs;
3. Evaluate the impact on air space and energy use of a large scale take-up of UAVs for medical logistics across the Solent region;
4. Understand stakeholder concerns about UAVs;
5. Understand the regulatory and governance needs associated with UAV interventions that will lead to energy benefits in logistics.

ELIGIBILITY:
Inclusion Criteria:

* Work Package 1

  * Task 1.1: key informants in appropriate job roles, with attention purposefully paid to gender and age balance of participants.
  * Task 1.2: Interviews - a purposeful recruitment strategy will seek participants with a range of socio-demographic characteristics. Questionnaire - Prolific (or a similar commercial company) will distribute the questionnaire (n~1000) to achieve a representative sample of the UK population.
  * Task 1.3: key informants in appropriate job roles, with attention purposefully paid to gender and age balance of participants.
* Work Package 5

  • Stakeholders with an interest in UAV use with a purposeful selection of participants with a range of socio-demographic characteristics.
* Work Package 6 • Anyone interacting with the serious game in dissemination events.

Exclusion Criteria:

• There are no specific exclusion criteria, though clearly some tasks require key informants with specific knowledge.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Task 1.1 - health staff/managers dealing with dispatch or receipt of patient diagnostics, bloods or pharmacy products at hospitals and GP surgeries, and transport staff..
  * Task 1.2 qualitative - key stakeholder groups involved in the project including, NHS staff, will be via the project teams' commercial partners, and the general public.
  * Task 1.2 quantitative - a representative sample of the UK population.
  * Task 1.3 - logistics staff and health staff/managers dealing with dispatch or receipt of patient diagnostics, bloods or pharmacy products at hospitals and GP surgeries.
  * Task 5.1 - key stakeholder groups involved in the project logistics providers, and a wider sample of the 144 organisations that responded to the Government consultation on the Future of Drones (January 2019).
  * Tasks 5.2 - Two sub-samples from task 5.1.
  * Task 6.2 - key stakeholders and members of the general public.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire to a representative panel of the public | 1 - 33 months
  To explore representations of UAVs
Questionnaire to a representative panel of the public | 1 - 33 months
  To understand public concerns
Questionnaire to a representative panel of the public | 1 - 33 months
  To determine how UAVs empower or constrain pathways to adoption

CONTACTS AND LOCATIONS:
Overall Officials: Janet Dickinson, Professor, Principal Investigator — Professor in Tourism
Locations (4):
- United Kingdom (4):
  - Dorset County Hospital NHS Foundation Trust, Dorchester, Dorset
  - University Hospitals Dorset NHS Foundation Trust, Poole, Dorset
  - Portsmouth Hospitals University National Health Service Trust, Portsmouth, Hampshire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire